CLINICAL TRIAL: NCT02293915
Title: Phase III Study of Sodium Oligo-mannurarate (GV-971) Capsule on Mild to Moderate Alzheimer Disease
Brief Title: An Efficacy and Safety Study of Sodium Oligo-mannurarate (GV-971) Capsule for the Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Greenvalley Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 971-III
Record Dates: First submitted 2014-11-13; First posted 2014-11-19 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Mild to Moderate Alzheimer Disease; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — GV-971

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sodium oligo-mannurarate 900mg (Experimental)
  Interventions: Drug: Sodium oligo-mannurarate 900mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium oligo-mannurarate 900mg — sodium oligo-mannurarate capsule 900mg twice a day for 24 weeks
  Other Names: GV-971
  Arms: sodium oligo-mannurarate 900mg
Drug: Placebo — simulant of sodium oligo-mannurarate capsule
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of Sodium Oligo-mannurarate (GV-971) in 36-week treatment of mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50-85 years (inclusive), no gender limitation;
2. Female subjects should be postmenopausal women (menopause >24 weeks), surgically sterilized women or women of child bearing age who agree to take effective contraceptive measures during the trial. Women of child bearing age and women less than 24 weeks from menopause must undergo urine pregnancy test in screening period and result must be negative;
3. Subjects have received education in primary school and above and are able to complete protocol specified cognitive ability test and other tests;
4. Impaired memory for at least 12 months, with a tendency of progressive aggravation;
5. Meet diagnostic criteria of probable AD according to National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) (1984);
6. Patients with mild to moderate disease, i.e. 11 ≤total MMSE score ≤26 (for subjects with primary school education, 11 ≤total MMSE score ≤22);
7. Total Hachinski Ischemia Scale (HIS) score ≤4 ;
8. Total Hamilton Depression Scale/17-item (HAMD) score ≤10;
9. In screening, cranial MRI plain scan and oblique coronal hippocampus scan must be performed, lacunar infarction lesions with a diameter larger than 2 cm ≤2, without lacunar infarction lesion in vital sites, such as thalamus, hippocampus, entorhinal cortex, paraolfactory cortex, cortex and other subcortical gray matter nuclei; MRI shows highest possibility of Alzheimer's disease (medial temporal lobe atrophy visual rating scale MTA grade ≥2);
10. Neurological examination shows no significant sign;
11. Subjects should have stable, reliable caregivers, or at least have frequent contact with caregivers (at least 4 days every week, at least 2 h every day), and caregivers will help patients in participation in this study. Caregivers must accompany subjects to participate in study visits and have sufficient interaction and communication with subjects, so as to provide valuable information on NPI, ADCS-ADL, CIBIC-plus scales.
12. Before implementation of any protocol related procedure or examination, subjects must sign the written informed consent form. If subjects can not sign due to limited cognition, legal guardians should sign on behalf of subjects and meanwhile, legal guardians should also sign the informed consent form.

Exclusion Criteria:

1. Participate in another clinical trial within 30 days prior to initiation of this study;
2. Pregnant or nursing women;
3. Dementia due to other causes: vascular dementia, central nervous system infection (e.g. AIDS, syphilis), Creutzfeldt-Jakob disease, Huntington's chorea, Parkinson's disease, dementia with Lewy bodies, traumatic dementia, other physical and chemical factors (e.g. drug poisoning, alcoholism, carbon monoxide poisoning), significant physical illness (e.g. hepatic encephalopathy, pulmonary encephalopathy), intracranial occupying lesion (e.g. subdural hematoma, brain tumor), endocrine disorders (e.g. thyroid disease, parathyroid disease) and dementia caused by vitamin or other factors;
4. Previous nervous system disorders (including stroke, optic neuromyelitis, Parkinson's disease, epilepsy);
5. Abnormal laboratory values: liver function (ALT, AST) > 1.5 times of upper limit of normal, Cr > 1.5 times of upper limit of normal, white blood cell count, platelet, hemoglobin below the lower limit of normal, blood glucose >1.5 times of upper limit of normal;
6. In screening, systolic blood pressure ≥160 mmHg or <90 mmHg, or diastolic blood pressure ≥100 mmHg or <60 mmHg;
7. Unstable or severe cardiac, pulmonary, hepatic, renal or hematopoietic disease (including unstable angina, uncontrolled asthma, active gastric bleeding and cancer), after 10 min rest, resting heart rate <55 bpm;
8. Visual or hearing disorder, preventing completion of neuropsychological test and scale evaluation;
9. In screening, MRI examination shows significant focal lesions, more than 2 lacunar infarction lesions with a diameter >2 cm, lacunar infarction lesions in vital sites, such as thalamus, hippocampus, entorhinal cortex, paraolfactory cortex, cortex and other subcortical gray matter nuclei; Fazekas scale for white matter lesions at ≥ grade 3;
10. Alcohol abuse or drug abuse;
11. Patients with psychosis, including severe depression;
12. Patients who are using drugs for Alzheimer's disease which can not be stopped;
13. Use of heparin, Propylene Glycol Mannurate Sulfate or Alginric Sodium Diester within 3 weeks prior to screening;
14. Inability to take trial drugs according to prescription, previous non-compliance with prescription or possibility of non-compliance with study treatment in the trial;
15. Investigators consider subjects can not complete this study;
16. Subjects in the phase II trial of the study drug;
17. Subjects are investigators participating in this study or their direct relatives, staff of Quintiles (Shanghai) or Shanghai Greenvalley Pharmaceutical Co., Ltd. or their direct relatives.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Improvement of Alzheimer's Disease Assessment Scale-cognitive subscale(ADAS-cog)/12 of sodium oligo-mannurarate capsule | 36 weeks

SECONDARY OUTCOMES:
Improvement of Clinician's Interview-Based Impression of Change Plus(CIBIC-plus) of sodium oligo-mannurarate capsule | 36 weeks
Improvement of Alzheimer's Disease Cooperative Study/Activities of Daily(ADCS-ADL) of sodium oligo-mannurarate capsule | 36 weeks
Improvement of Neuropsychiatric Inventory(NPI) of sodium oligo-mannurarate capsule | 36 weeks
Glucose metabolism of bilateral temporoparietal cortex | 36 weeks
  Obtained by Positron Emission Tomography in two sites.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Beijing, Beijing, Beijing Municipality
  - Chongqing, Chongqing, Chongqing Municipality
  - Fujian, Fuzhou, Fujian
  - Guangzhou, Guangzhou, Guangdong
  - Wuhan, Wuhan, Hubei
  - Changsha, Changsha, Hunan
  - Nanjing, Nanjing, Jiangsu
  - Suzhou, Suzhou, Jiangsu
  - Yangzhou, Yangzhou, Jiangsu
  - Jinan, Jinan, Shandong
  - Shanghai, Shanghai, Shanghai Municipality
  - Xi'an, Xi’an, Shanxi
  - Sichuan, Chengdu, Sichuan
  - Tianjin, Tianjin, Tianjin Municipality
  - Hangzhou, Hangzhou, Zhejiang
  - Wenzhou, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrari C, Sorbi S. The complexity of Alzheimer's disease: an evolving puzzle. Physiol Rev. 2021 Jul 1;101(3):1047-1081. doi: 10.1152/physrev.00015.2020. Epub 2021 Jan 21. PMID 33475022